CLINICAL TRIAL: NCT01385501
Title: Educational Intervention to Improve Vaccine Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Elizabeth Williams, Research Instructor, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VA 1111
Record Dates: First submitted 2011-03-02; First posted 2011-06-30 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Vaccine Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- routine care (No Intervention)
- Educational intervention group (Experimental)
  Interventions: Other: Video intervention along with educational hand out

INTERVENTIONS:
Other: Video intervention along with educational hand out — The interventional group will be shown an 8 minute video addressing common concerns of vaccine hesitant parents. Then, they will be provided with a handout describing how to find accurate vaccine information on the internet and a handout on more common questions from vaccine hesitant parents.
  Arms: Educational intervention group

SUMMARY:
This research project will develop an educational intervention to improve immunization acceptance by vaccine hesitant parents. This is prospective interventional case-control trial, where the investigators will provide the intervention in the clinical setting. Enrollees will be screened and selected if they meet criteria for "vaccine hesitancy". The investigators will conduct follow up surveys following the intervention to assess change in attitude and follow immunization rates through 18 month well visit.

DETAILED DESCRIPTION:
The intervention is a 8 minute video addressing common concerns that have been reported by vaccine hesitant parents. The video includes an expert in pediatric infectious diseases answering these common questions as well as 3 parental accounts of children who contracted vaccine preventable diseases. Also, the interventional group will be provided with two handouts: one listed information on how parents can find accurate vaccine information on the internet, and another that addresses more common concerns of vaccine hesitant parents and available for our use from the Children's Hospital of Philadelphia Vaccine Center website.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old for parent
* < 30 days old for infant
* full term (>37 weeks gestational age) infant

Exclusion Criteria:

* none

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in parental attitude regarding vaccines | 6-8 weeks
  Parental attitudes regarding vaccines will be assessed upon screening to determine the parental level of hesitancy regarding childhood vaccines. We will will use the same survey questions again immediately after the intervention and at the 2 month visit to measure change in parental attitude. We will also survey the control group at the 2 month check as well to compare attitude change without the intervention.

SECONDARY OUTCOMES:
Vaccination rates of control and interventional groups | 6-8 weeks, 19 months
  Vaccination rates will be compared between groups at both 2 months of age and 19 months of age.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Franklin Pediatric Associates, Franklin, Tennessee
  - University Pediatrics, Nashville, Tennessee